CLINICAL TRIAL: NCT00637598
Title: Early Detection of Breast Cancer Using Tomosynthesis Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00013552; 6024 (Other: DUMC Eirb:Pro00013552); 6503 (Other: Duke legacy protocol ID)
Record Dates: First submitted 2008-03-12; First posted 2008-03-18 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2014-07

CONDITIONS: Breast Neoplasms
Keywords: Diagnostic Imaging; Mammography; Breast Tomosynthesis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tomosynthesis scans (Experimental): This is a case-only study with only one group/cohort. All women receive both mammography and tomosynthesis imaging.
  Interventions: Radiation: Mammography and tomosynthesis imaging

INTERVENTIONS:
Radiation: Mammography and tomosynthesis imaging — All subjects receive the same radiation dose associated with mammography and tomosynthesis imaging (which is comparable to mammography).
  Other Names: Digital breast tomosynthesis (DBT); Breast tomosynthesis; full field digital mammography (FFDM); screen-film mammography; film-screen mammography

SUMMARY:
The purpose is to develop digital tomosynthesis to improve the detection of breast cancers. The aims are optimizing digital mammography and tomosynthesis acquisition, creating visualization tools, prospective pilot studies to evaluate radiologist performance, and computer-aided detection.

DETAILED DESCRIPTION:
Finding breast cancer early has been shown to improve the chance of survival. Mammography (x-ray imaging of the breast) helps find breast cancer early. Some breast cancers, however, are not seen on mammography, which creates two-dimensional images for the radiologist to see. The goal of this study is to make a breast tomosynthesis or tomosynthesis 3D (three-dimensional) x-ray system by taking x-ray images from many angles. This is similar to a CAT (computerized axial tomography) scan for the breast and can give radiologists 3D information so that they can find breast cancers which might otherwise be hidden from view.

ELIGIBILITY:
Inclusion Criteria:

All Subjects accepted for this clinical study must:

* Be already scheduled to undergo screening mammography, diagnostic mammography, or breast biopsy for standard clinical indications
* Provide written informed consent
* Be able to communicate effectively with clinical study personnel.

Exclusion Criteria:

Subjects with any of the following conditions will be excluded from this clinical study:

* Childbearing potential and subject refuses serum pregnancy test or test result is positive.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2004-11; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Radiologist ROC (receiver operating characteristic) area under curve (AUC) | at imaging review by the end of the study, approximately 9 years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Y Lo, PhD, Principal Investigator — Duke Health
Locations (1):
- DUMC Mammography, Duke South Hospital, 2nd floor, Durham, North Carolina, United States